CLINICAL TRIAL: NCT06455956
Title: New Potential Biomarkers for Diagnosis of Growth Hormone (GH) Deficiency and Early Assessment of Response to GH Treatment for Appropriate Personalization of Therapy
Brief Title: Use of miRNAs in Growth Hormone Deficiency (GHD)
Acronym: GH-miRNA2
Status: Recruiting | Type: Observational
Sponsor: University of Parma (Other)
Collaborators: Azienda Ospedaliera Universitaria Policlinico "G. Martino" (Other); Ospedali Riuniti Ancona (Other); Federico II University (Other); Azienda Unita Sanitaria Locale di Piacenza (Other); Azienda Ospedaliero Universitaria Policlinico Modena (Other); Azienda USL Reggio Emilia - IRCCS (Other Government); Azienda Ospedaliero-Universitaria Consorziale Policlinico di Bari (Other); Ospedali Riuniti di Foggia (Other); IRCCS Ospedale San Raffaele (Other); Università degli Studi del Piemonte Orientale Amedeo Avogadro (Other); IRCCS Azienda Ospedaliero-Universitaria di Bologna (Other); Istituto Auxologico Italiano (Other); OSPEDALE CARLO POMA ASST MANTOVA (Unknown); University of Campania Luigi Vanvitelli (Other); Fondazione IRCCS Ca' Granda, Ospedale Maggiore Policlinico (Other)
Responsible Party: Sponsor
Other Study IDs: 821/2022/OSS/UNIPR
Record Dates: First submitted 2024-06-06; First posted 2024-06-13 (Actual); Last update posted 2024-06-13 (Actual); Status verified 2024-05

CONDITIONS: Growth Hormone Deficiency
Keywords: growth hormone; miRNA; growth hormone deficiency; growth hormone treatment; small for gestational age; Turner syndrome; Noonan syndrome; SHOX deficiency
MeSH Terms: conditions — Dwarfism, Pituitary; Turner Syndrome; Noonan Syndrome

STUDY DESIGN:
Observational Model: Cohort | Time Perspective: Prospective
Biospecimen Retention: Samples Without DNA — Serum
Oversight: FDA-regulated Drug: No | FDA-regulated Device: No

SUMMARY:
This study aims at improving knowledge about the diagnosis of growth hormone deficiency (GHD) and treatment with growth hormone (GH), with the goal of providing information on the presence of new biomarkers, such as miRNAs, for diagnostic and therapeutic purposes, with the goal of establishing a personalized GH treatment scheme, optimizing resources, reducing costs, and improving outcomes.

DETAILED DESCRIPTION:
In 200 prepubertal and pubertal subjects with the suspicion of GHD, the levels of three specific circulating miRNas will be measured to establish whether they can be used for the diagnosis of GH deficiency. In subjects with isolated idiopathic GHD (IIGHD), short statured patients born SGA, Noonan and Turner syndromes, and SHOX deficiency, we will also assess the changes of the identified miRNAs before and after 3 months on GH therapy to verify an early growth prediction model for growth response at 12 months on treatment. Finally, we plan to identify any differences in these miRNAs at 3 months on treatment using daily GH versus weekly (long-acting) GH.

ELIGIBILITY:
Inclusion Criteria for aim 1:

* Children with short stature and suspicion of GHD
* Subjects with organic GH deficiency

Exclusion criteria for aim 1:

-Subjects with underlying genetic conditions and chronic diseases

Inclusion Criteria for aim 2-3-5:

* patients having confirmed GHD enrolled for aim 1
* patients with growth failure and born SGA (>4 yr of age)
* patients with Noonan and Turner syndrome and growth failure
* patients with short stature homeobox-containing gene deficiency (SHOXD) and growth failure

Inclusion Criteria for aim 4:

- Isolated idiopathic prepubertal naive GHD subjects on long-acting versus daily GH therapy

Ages: 2 Years to 15 Years | Sex: All | Healthy Volunteers: No
Age Groups: Child
Study Population: All patients will be investigated in routine practice during the normal workup for short stature and stunted growth. Treatment will be also delivered accordind to standard care indications and as established by regulatory agencies in Italy.
Sampling Method: Non-Probability Sample
Enrollment: 400 (Estimated)
Dates: Start 2023-04-13 (Actual); Primary Completion 2025-03-31 (Estimated); Study Completion 2026-03-01 (Estimated)

PRIMARY OUTCOMES:
Assessing new biomarkers for the diagnosis of GHD | 3 years
  The 1st objective will consist in the enrolment of 200 subjects, nationwide, undergoing standard routine work-up for the diagnosis of GHD. The specific miRNAs will be measured at the time of both stimulation tests in order to include subjects with both confirmed and unconfirmed GHD and guarantee reproducibility; in addition, subjects with organic GH deficiency will be included.
Measuring miRNA changes after 3 months on GH therapy | 3 years
  The 2nd objective will consist in measuring these specific miRNAs before and at 3 months on treatment in 200 subjects with isolated idiopathic GHD(IIGHD), and in 60 short statured patients born SGA, in 60 having Noonan and Turner syndromes, and in 30 with SHOX deficiency, according to current indications to verify whether changes are confirmed in pubertal versus prepubertal subjects and in conditions other than IIGHD.
Multiple linear regression models | 3 years
  The 3rd objective will consist in investigating the major determinants of height variations between 0 and 6 months, 0 and 12 months and the variance of growth rate variation between 0 and 6 months including the levels and/or changes in the specific miRNAs at baseline and at 3 months on treatment by using multiple linear regression models to establish early prediction models of growth response..
Measuring miRNA changes between daily and long-acting GH therapy | 3 years
  The 4th objective will consist in measuring these specific miRNAs before and at 3 months on treatment in children with IIGHD being treated with daily versus longacting GH. Findings will be compared with those in the IIGHD group receiving daily GH treatment as an exploratory task, thus, only a small number of subjects will be enrolled, and anyway as many as possible.

SECONDARY OUTCOMES:
Sex-specific miRNA changes after 3 months on long-acting GH therapy | 3 years
  Any differences between males and females in miRNAs expression after 3 months of long-acting GH therapy will be evaluated.

CONTACTS AND LOCATIONS:
Overall Officials: Maria E Street, MD, PhD, Principal Investigator — University of Parma
Locations (1):
- University of Parma, Parma, Emilia-Romagna, Italy

IPD SHARING:
Plan to Share IPD: No